CLINICAL TRIAL: NCT01083667
Title: Phase I/II Study of SOD1 Inhibition by Pyrimethamine in Familial ALS
Brief Title: SOD1 Inhibition by Pyrimethamine in Familial Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Muscular Dystrophy Association (Other)
Responsible Party: Principal Investigator, Dr. Dale J. Lange, Neurologist in Chief, Weill Medical College of Cornell University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0903010259
Record Dates: First submitted 2009-12-17; First posted 2010-03-10 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-05

CONDITIONS: Familial Amyotrophic Lateral Sclerosis
Keywords: ALS; Familial ALS; SOD1 Gene Mutation
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Pyrimethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pyrimethamine (Experimental): Open label. Only one arm will receive the intervention.
  Interventions: Drug: Pyrimethamine

INTERVENTIONS:
Drug: Pyrimethamine — Open Label, dose escalating,
  Other Names: Daraprim

SUMMARY:
The objective of this study will be to evaluate the safety, tolerability and effect on SOD1 levels by pyrimethamine in patients with familial amyotrophic lateral sclerosis.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a neurodegenerative disease causing relentlessly progressive weakness of the arms, legs and respiratory muscles that is uniformly fatal. There are approximately 30,000 patients living with ALS in the United States. There is no treatment. The cause is uncertain in most patients. However, 3% of patients (< 1000 in number) have a familial form of ALS (FALS), phenotypically identical to the sporadic illness, that is caused by a mutation in the gene coding for the free radical scavenging enzyme copper/zinc superoxide dismutase (SOD1). Inserting the SOD1 mutant gene into mice causes them to develop a disease closely resembling ALS.

Inhibiting expression of the SOD1 gene prevents animals from developing the disease. Increasing or decreasing the number of mutated genes proportionately speeds or slows the progression of the disease. Therefore, reducing SOD1 levels in patients with SOD1 associated FALS may be a promising therapeutic approach. Through an extensive in vitro screening program for medications having the ability to reduce SOD1 levels, several molecules that reduce SOD1 protein levels are known. One of the most potent molecules is pyrimethamine, an FDA approved medication used for the treatment of malaria and toxoplasmosis. Pyrimethamine dramatically reduces SOD1 levels in mice and our preliminary studies show similar findings in humans. Our study's primary objective is to determine if familial ALS patients taking pyrimethamine will show a decline in SOD1 levels in the CSF by 15% or more. We will also determine if SOD1 and pyrimethamine are present in the blood and if the SOD-1 levels decline over the course of the study. We will also evaluate the safety and tolerability of pyrimethamine in patients with FALS. Secondary objectives will be to determine dose optimization for maximal SOD1 level reduction and tolerability of medication. We will also assess the feasibility of proceeding to phase II/III studies using pyrimethamine. Change in ALS-FRS, Appel ALS score and quality of life will also be measured. A clinical effect realized in patients with FALS associated with an SOD1 mutation may serve as an important foundation toward finding a treatment for sporadic ALS.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with definite, probable, or laboratory supported probable ALS will be eligible.

  1. ALS diagnosed as probable, laboratory supported probable or definite according to the World Federation of Neurology El Escorial criteria [Brooks et al. 2000]
  2. Age 18 or older
  3. Capable of providing informed consent and complying with trial procedures
  4. SOD1 mutation confirmation by study team
  5. Not taking Riluzole (Rilutek) or on a stable dose for 30 days
  6. Not taking Coenzyme QR10R or on a stable dose and brand for 30 days
  7. Absence of exclusion criteria

Exclusion Criteria:

1. History or evidence of malabsorption syndromes
2. Exposure to any experimental agent within 30 days of onset of this protocol
3. Women who are pregnant or planning to become pregnant
4. Women of childbearing potential not practicing contraception
5. Women who are breastfeeding
6. Enrollment in another research study within 30 days of or during this trial
7. Alcoholism
8. Patients taking phenytoin (Dilantin) or other therapy affecting folate levels
9. Dementia (MMSE <22)
10. Seizure disorder
11. Folate deficiency
12. Megaloblastic anemia
13. Cardiovascular disorder/arrhythmia
14. Impaired kidney function, defined as creatinine levels of 2.5 x ULN
15. Impaired liver function, defined as AST or ALT of 3 X ULN
16. Advanced ALS patients, defined as those with any of the following: forced vital capacity <60% (use of BIPAP is allowed); tracheostomy; or mechanical ventilation
17. Use of any of the following medications: cytosine, arabinoside, methotrexate, daunorubicin, sulfonamides, zidovudine, lorazepam, coumadin, sulfamethoxazole, and trimethoprim
18. Patients taking Lithium within 30 days of or during this trial
19. Incapable of providing informed consent and complying with trial procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-11; Primary Completion 2014-12 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dale J. Lange, M.D., Principal Investigator — Hospital for Special Surgery/Weill Cornell Medical Center
Locations (5):
- United States (2):
  - Weill Cornell Medical Center/New York Presbyterian Hospital, New York, New York
  - Methodist Neurological Institute, Houston, Texas
- Universitäts- und Rehabilitationskliniken Ulm, Ulm, Germany
- Milano Neurological Institute, Milan, Italy
- Umea University, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient were recruited from all sites and referrals received from other physicians. Subjects also contacted sites from ClinicalTrials.gov posting
Period: Overall Study
Arm/Group | Pyrimethamine
Started | 32 (enrolled)
Completed | 22 (22 completed to visit 9, the last visit on study.)
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Pyrimethamine
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants] — age of subjects enrolled
  Participants
    <=18 years | 0
    Between 18 and 65 years | 31
    >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 48 [19 to 72]
Sex: Female, Male [Count of Participants; unit: Participants] — gender of subjects enrolled
  Participants
    Female | 16
    Male | 16
Region of Enrollment [Number; unit: participants] — enrollment of subjects in US and Europe
  participants
    United States | 20
    Italy | 8
    Germany | 4

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in SOD1 CSF
Description: Reported change in mean SOD1 CSf from baseline to visit 6 (week 18) and end of study for all subjects who completed the measure
Time Frame: baseline, Visit 6 week 18, end of study
Population: 24 subjects completed up to visit 6 and 21 subjects for final study visit. Reported is the change in SOD1 CSF from baseline to week 36.
Measure: Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Pyrimethamine
Number analyzed (Participants) | 22
ng/ml | 6.8 [3.4 to 10.3]

2. Secondary Outcome: Appel ALS Score
Description: an objective and timed measurement of strength and function of subjects including muscle testing, respiratory function and fine motor function, all summed together for a total value, and is measured at baseline, visit 2, visit 6 and end of study. The scale ranges from 30 in a healthy person to to 164 in a maximally impaired person; an increase in score indicates progression and is expected in disease progression.
Time Frame: Week 0, 6, 18, and end of study
Population: 22 subjects completed to visit 9 and had a final score for Appel Score. Reported is the mean change from Baseline to week 36
Measure: Number (95% Confidence Interval); unit: units on a scale
Arm/Group | Pyrimethamine
Number analyzed (Participants) | 22
units on a scale | 18 [12 to 24]

ADVERSE EVENTS:
Time Frame: AE's were collected over the course of the study and up to 30 days following the last dose taken.
Description: CTCAE version 4.0 was used to assess the severity of AE's experienced during the study. This uses a grading system (referring to the severity) to assess the AEs. The CTCAE v4.0 displays Grades 1-5 with unique clinical descriptions of severity for each AE based on this general guideline: G1 Mild AE, G2 Moderate AE, G3 Severe or medically significant but not immediately life-threatening, G4 Life-threatening, G5 Death related to AE.
  SAE reporting per criteria od clinicaltrials.gov
Arm/Group | Pyrimethamine
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 1/32
Other Adverse Events (participants affected / at risk) | 14/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pyrimethamine (N=32)
Pneumonia (Infections and infestations) | 1 (1) — Patient admitted to the hospital with pneumonia while on study, course complicated by discovery of a congenital esophageal fistula which was repaired, patient discharged home and continued on the study. The event was not related to study medication.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pyrimethamine (N=32)
Headache (Nervous system disorders) | 13 (13) — headache following spinal tap
Nausea (Metabolism and nutrition disorders) | 14 (14) — GI nausea
Diarrhea (Metabolism and nutrition disorders) | 6 (6)
Pain (Musculoskeletal and connective tissue disorders) | 5 (5) — Pain following Spinal Tap
weight loss (Metabolism and nutrition disorders) | 3 (3) — greater than 5% was recorded
Upper respiratory infection (Infections and infestations) | 4 (4) — URI infection and Pneumonia
decreased appetite (Metabolism and nutrition disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No